CLINICAL TRIAL: NCT00867789
Title: Trimethoprim-sulfamethoxazole Versus Placebo in the Treatment of Cutaneous Abscesses in the Emergency Department
Brief Title: Antibiotics Versus Placebo in the Treatment of Abscesses in the Emergency Department
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment due to subjects not meeting inclusion/exclusion criteria
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Blue Cross Blue Shield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0810-162
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Abscess
Keywords: abscess; outcomes; antibiotics; incision and drainage; skin abscess
MeSH Terms: conditions — Abscess; Surgical Wound | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trimethoprim-sulfamethaxazole (Experimental): Incision and drainage of the abscess and treatment with oral TMP-SMX (100 patients)
  Interventions: Drug: Trimethoprim-sulfamethoxazole
- Sugar pill (Placebo Comparator): Incision and drainage of the abscess and treatment with oral placebo (100 patients)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Trimethoprim-sulfamethoxazole — 10mg/kg/day (based on trimethoprim component), divided twice daily for ten days (maximum dose: 160mg (TMP component) per dose)
  Other Names: Bactrim
  Arms: Trimethoprim-sulfamethaxazole
Drug: Sugar pill — 10mg/kg/day divided twice daily for ten days. Placebo liquid will contain simple syrup, lactose powder, grape flavor, and food coloring. Placebo capsules will contain lactose powder.
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine if there is a difference between an antibiotic, trimethoprim-sulfamethoxazole versus placebo in healing outcomes of soft tissue abscesses following incision and drainage.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 months to 17 years
* Single, localized soft tissue abscesses requiring incision and drainage with purulent material obtained
* Diameter of the abscess less than 5cm as measured by the treating physician

Exclusion Criteria:

* Signs of systemic illness or ill-appearing, as determined by the treating physician
* Admission to the hospital following treatment in the Emergency Department
* Known sulfa allergy
* Immunocompromised patients
* Soft tissue abscesses involving the perineum (labia, scrotum, penis, perirectal)
* Previous antibiotic use (for any reason) in the past seven days
* Non-English speaking patients and families

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Giovanni, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Background] McCaig LF, McDonald LC, Mandal S, Jernigan DB. Staphylococcus aureus-associated skin and soft tissue infections in ambulatory care. Emerg Infect Dis. 2006 Nov;12(11):1715-23. doi: 10.3201/eid1211.060190. PMID 17283622
- [Background] Halvorson GD, Halvorson JE, Iserson KV. Abscess incision and drainage in the emergency department--Part I. J Emerg Med. 1985;3(3):227-32. doi: 10.1016/0736-4679(85)90077-0. PMID 4093575
- [Background] Meislin HW, McGehee MD, Rosen P. Management and microbiology of cutaneous abscesses. JACEP. 1978 May;7(5):186-91. doi: 10.1016/s0361-1124(78)80097-5. PMID 349218
- [Background] Macfie J, Harvey J. The treatment of acute superficial abscesses: a prospective clinical trial. Br J Surg. 1977 Apr;64(4):264-6. doi: 10.1002/bjs.1800640410. PMID 322789
- [Background] Burney RE. Incision and drainage procedures: soft tissue abscesses in the emergency service. Emerg Med Clin North Am. 1986 Aug;4(3):527-42. No abstract available. PMID 3720656
- [Background] Llera JL, Levy RC, Staneck JL. Cutaneous abscesses: natural history and management in an outpatient facility. J Emerg Med. 1984;1(6):489-93. doi: 10.1016/0736-4679(84)90002-7. PMID 6444142
- [Background] Llera JL, Levy RC. Treatment of cutaneous abscess: a double-blind clinical study. Ann Emerg Med. 1985 Jan;14(1):15-9. doi: 10.1016/s0196-0644(85)80727-7. PMID 3880635
- [Background] Frank AL, Marcinak JF, Mangat PD, Tjhio JT, Kelkar S, Schreckenberger PC, Quinn JP. Clindamycin treatment of methicillin-resistant Staphylococcus aureus infections in children. Pediatr Infect Dis J. 2002 Jun;21(6):530-4. doi: 10.1097/00006454-200206000-00010. PMID 12182377
- [Background] Frank AL, Marcinak JF, Mangat PD, Schreckenberger PC. Community-acquired and clindamycin-susceptible methicillin-resistant Staphylococcus aureus in children. Pediatr Infect Dis J. 1999 Nov;18(11):993-1000. doi: 10.1097/00006454-199911000-00012. PMID 10571437
- [Background] Frazee BW, Lynn J, Charlebois ED, Lambert L, Lowery D, Perdreau-Remington F. High prevalence of methicillin-resistant Staphylococcus aureus in emergency department skin and soft tissue infections. Ann Emerg Med. 2005 Mar;45(3):311-20. doi: 10.1016/j.annemergmed.2004.10.011. PMID 15726056
- [Background] Mishaan AM, Mason EO Jr, Martinez-Aguilar G, Hammerman W, Propst JJ, Lupski JR, Stankiewicz P, Kaplan SL, Hulten K. Emergence of a predominant clone of community-acquired Staphylococcus aureus among children in Houston, Texas. Pediatr Infect Dis J. 2005 Mar;24(3):201-6. doi: 10.1097/01.inf.0000151107.29132.70. PMID 15750454
- [Background] Fergie JE, Purcell K. Community-acquired methicillin-resistant Staphylococcus aureus infections in south Texas children. Pediatr Infect Dis J. 2001 Sep;20(9):860-3. doi: 10.1097/00006454-200109000-00007. PMID 11734764
- [Background] Sattler CA, Mason EO Jr, Kaplan SL. Prospective comparison of risk factors and demographic and clinical characteristics of community-acquired, methicillin-resistant versus methicillin-susceptible Staphylococcus aureus infection in children. Pediatr Infect Dis J. 2002 Oct;21(10):910-7. doi: 10.1097/00006454-200210000-00005. PMID 12394811
- [Background] Purcell K, Fergie J. Epidemic of community-acquired methicillin-resistant Staphylococcus aureus infections: a 14-year study at Driscoll Children's Hospital. Arch Pediatr Adolesc Med. 2005 Oct;159(10):980-5. doi: 10.1001/archpedi.159.10.980. PMID 16203945
- [Background] Kaplan SL. Treatment of community-associated methicillin-resistant Staphylococcus aureus infections. Pediatr Infect Dis J. 2005 May;24(5):457-8. doi: 10.1097/01.inf.0000164162.00163.9d. No abstract available. PMID 15876948
- [Background] Gonzalez BE, Martinez-Aguilar G, Hulten KG, Hammerman WA, Coss-Bu J, Avalos-Mishaan A, Mason EO Jr, Kaplan SL. Severe Staphylococcal sepsis in adolescents in the era of community-acquired methicillin-resistant Staphylococcus aureus. Pediatrics. 2005 Mar;115(3):642-8. doi: 10.1542/peds.2004-2300. PMID 15741366
- [Background] Klevens RM, Morrison MA, Nadle J, Petit S, Gershman K, Ray S, Harrison LH, Lynfield R, Dumyati G, Townes JM, Craig AS, Zell ER, Fosheim GE, McDougal LK, Carey RB, Fridkin SK; Active Bacterial Core surveillance (ABCs) MRSA Investigators. Invasive methicillin-resistant Staphylococcus aureus infections in the United States. JAMA. 2007 Oct 17;298(15):1763-71. doi: 10.1001/jama.298.15.1763. PMID 17940231
- [Background] Lee MC, Rios AM, Aten MF, Mejias A, Cavuoti D, McCracken GH Jr, Hardy RD. Management and outcome of children with skin and soft tissue abscesses caused by community-acquired methicillin-resistant Staphylococcus aureus. Pediatr Infect Dis J. 2004 Feb;23(2):123-7. doi: 10.1097/01.inf.0000109288.06912.21. PMID 14872177

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trimethoprim-sulfamethaxazole | Sugar Pill
Started | 70 | 70
Completed | 68 | 70
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trimethoprim-sulfamethaxazole | Sugar Pill | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 70 | 70 | 140
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 32 | 30 | 62
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Health Outcomes After Use With Trimethoprim-sulfamethaxazole
Time Frame: two years
Measure: Number; unit: Percentage of outcomes assessed
Arm/Group | Trimethoprim-sulfamethaxazole | Sugar Pill
Number analyzed (Participants) | 70 | 70
Percentage of outcomes assessed | 0 | 0

ADVERSE EVENTS:
Arm/Group | Trimethoprim-sulfamethaxazole | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No